CLINICAL TRIAL: NCT02827019
Title: Newborn in Helathy Birthroom: Assessment of Pratical Home and Mother Lived
Acronym: EPAVM
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EPAVM
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Newborns; Motherhood; Delivery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — a questionnaire made puerperium the 2nd day of life during the interview with the parents on the basis of a semi-structured interview about the progress of the birth and the immediate postpartum period using the memories of parents

SUMMARY:
Motherhood Our Lady of Good Help is from the 2006 merger of three hospitals, St. Joseph, Our Lady of Good Help and Saint-Michel. She was transferred to a new building in the heart of Paris Saint-Joseph Hospital Group website in March 2011. The premises of the birth room are spacious and nice. All delivery rooms are supposed to welcome the mother and child when the birth goes smoothly. There is a resuscitation room (called "Nursery") for newborns requiring medical care. But since the installation in the new building, the investigators had the impression that a number of children born without pathology futures and with good adaptation at birth passed through this room for no apparent medical reason.

The investigators wanted to make an inventory of home practice healthy newborns in our maternity, evaluate the reasons for a possible separation and appreciate the feelings of mothers cope with this separation.

DETAILED DESCRIPTION:
Objective of the study Evaluation of home practices of a healthy newborn in the delivery room: skin processing conditions skin, reasons for separation between mother and child and maternal felt appreciation.

Methodology :

DESIGN:

Study single-center observational descriptive, carried out over a period of 8 weeks during the months of January and February 2015 in the Maternity Our Lady of relief

Acquisition of data:

- From a survey conducted in puerperium the 2nd day of life during the interview with the parents on the basis of a semi-structured interview about the progress of the birth and the immediate postpartum period using memories of parents. The questionnaire included a section on skin to skin layout with the newborn (information on skin to skin, original maturity), the output or not the child of the delivery room (reason given, period of separation , felt the mother), the conditions of return (naked or dressed, delivered or not skin to skin, conditions the first feeding), the place of the first examination of the newborn and the overall satisfaction of the mother.

The reasons for the release of children were classified as routine care (weight, measurements, toilet or exam), clinical monitoring of the Child (declogging, monitoring of respiratory discomfort or poor adaptation), warming the child, simple or complicated maternal care) and implementation of a levy (gastric, Rh, pH). The traceability of the reason for leaving the newborn in the delivery room was searched in the newborn monitoring sheet (production of a levy, the child's warming, clinical monitoring of the child) and in the medical record of the mother (complicated birthing suites with uterus bleeding or tearing).

- And from the collection of the passage of newborns in the "nursery" of the delivery room of 11 days. The collection form was filled by the auxiliary of the delivery room should note that with each pass of a newborn in the "nursery", the time of birth, time of arrival and departure and the main reason for the passage of the newborn in the "nursery." The reasons were categorized (routine care, achieving a levy, the child's warming, clinical monitoring of the child, the mother care).

Analysis: This is primarily a descriptive analysis. A comprehensive description of the sample was carried out by giving the frequencies of different categories for qualitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Newborns at term (≥ 37 weeks of gestation), eutrophic (≥ 10th p)
* Born vaginally
* Good adaptation to extra-uterine life: breathe or scream, has good skin color, a good tone with an Apgar score ≥7
* Absence of meconium amniotic fluid

Exclusion Criteria:

* Preterm (<37 weeks of gestation), hypotrophe (<10th cp)
* Born by caesarean section
* Poor adaptation to extra-uterine life
* Amniotic fluid meconium

Ages: 1 Day to 11 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: mothers whose newborns meet the inclusion criteria. They are in good health before birth mothers in normal
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
Number of routine care | within the first 11 days life
  Will be considered as routine care: weighing, measurement, toilet or review

SECONDARY OUTCOMES:
Number of realization of a levy | within the first 11 days life
  for gastric fluid or blood
Number of times that the Child was warming | within the first 11 days life
Number of Clinical monitoring of the child | within the first 11 days life
Number of care provided to the mother | within the first 11 days life
  Number and description of care provided to the mother

CONTACTS AND LOCATIONS:
Overall Officials: TASSEAU Angelique, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France